CLINICAL TRIAL: NCT00239304
Title: A Phase I/II Trial of ZD1839 (Iressa) Given Concurrently With Cisplatin and Radiotherapy in Patients With Locally Advanced Head and Neck Cancer
Brief Title: Gefitinib (Iressa) in Combo With Chemoradiation in Patients With Locally Advanced Head & Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0151
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Head and Neck Neoplasms
Keywords: Stage III Head and Neck Cancer; Stage IV Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Gefitinib; Cisplatin; Radiotherapy

INTERVENTIONS:
Drug: Gefitinib
Drug: Cisplatin
Procedure: Radiotherapy

SUMMARY:
To determine the safety and tolerability of gefitinib in combination with cisplatin and radiation (3D-CRT or IMRT) in patients with locally advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed head and neck cancer
* Lymph node negative or positive
* Metastasis negative
* Chemo- and radiotherapy naïve
* WHO 0-2
* Measurable disease by RECIST
* Written informed consent

Exclusion Criteria:

* Severe alcohol abuse
* Active ILD
* Co-existing chronic gastrointestinal disease(s)
* Brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-06; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Parts 1 and 2: Safety (Incidence of DLTs)
Part 3: Safety and tolerability

SECONDARY OUTCOMES:
Parts 2 and 3: Efficacy (Incidence of complete response at 3 months after the end of trial treatment based on RECIST criteria)
Exploratory Outcome: EGFR-1 expression, amplification and activation Serum VEGF levels

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Finland Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Centre, Helsinki, Finland